CLINICAL TRIAL: NCT03271307
Title: Use of HIV Self-Test Kits to Increase Identification of HIV-Infected Individuals and Their Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Partners in Hope, Inc. (Industry); United States Agency for International Development (USAID) (U.S. Federal Agency); Right to Care (Other); Ministry of Health, Malawi (Other Government)
Responsible Party: Principal Investigator, Kathryn L. Dovel, PhD, Adjunct Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-000109
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections
Keywords: self-test; testing; cost-effectiveness
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: The study will include two arms and methodology: (Aim 1) A cluster-randomized trial comparing HIV testing strategies for OPD clients, clustered by health facility; and (Aim 2) A individual-randomized trial comparing HIV testing strategies for partners of HIV-positive clients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- AIm 1: Standard of care (No Intervention): Facilities assigned to the standard of care arm will receive no intervention and will continue with Ministry of Health National HIV Guidelines for provider-initiated testing and counseling (PITC) for outpatients in Aim 1. PITC guidelines recommend providers inform their OPD clients about HIV testing and refer them to HIV testing services at the facility.
- Aim 1: Optimized standard of care (Experimental): Facilities assigned to the optimized standard of care arm will receive additional guidance and support from the study team to adopt the Ministry of Health National HIV Guidelines for provider-initiated testing and counseling (PITC) for Aim 1.
  Interventions: Behavioral: Optimized PITC
- Aim 1: Facility HIVST (Experimental): Facilities assigned to the HIVST arm will implement HIVST procedures in lieu of recommendations provided by the Ministry of Health National HIV Guidelines (PITC).
  Interventions: Diagnostic Test: Facility HIVST
- Aim 2: Standard of care (No Intervention): Facilities assigned to the standard of care arm will receive no intervention and will continue with Ministry of Health National HIV Guidelines for index HIV testing for sexual partners of HIV-positive clients. Partner referral slips will be given to HIV-positive clients to encourage partner testing.
- Aim 2: Index HIVST (Experimental): Facilities assigned to the HIVST arm will implement HIVST procedures in lieu of recommendations provided by the Ministry of Health National HIV Guidelines (partner referral slips).
  Interventions: Diagnostic Test: Index HIVST

INTERVENTIONS:
Behavioral: Optimized PITC — Providers will receive training on the importance of HIV testing and their role in testing as part of OPD care and morning HIV testing will be offered. Providers will receive job aids on the importance of referring patients for HIV testing, and the study team will conduct regular monitoring and evaluation on PITC implementation.
  Other Names: Optimized standard of care
  Arms: Aim 1: Optimized standard of care
Diagnostic Test: Facility HIVST — HIVST will be carried out in a group setting among patients in the waiting area of OPD clinics. Eligible clients will receive education about HIV testing and a demonstration of how to use and interpret results of a self-test kit will occur in the group setting. Participants will use the HIVST kit in a group setting and will be given private settings (private room or booth) to interpret their results. Participants will disclose their results to their OPD provider if they choose. Routine linkage to confirmatory testing and ART initiation will be conducted.
  Arms: Aim 1: Facility HIVST
Diagnostic Test: Index HIVST — HIVST demonstration and distribution will be provided to HIV-positive clients in participating facilities to distribute to their partners. Partners who have a reactive HIVST test result, or are unable or unwilling to use HIVST, will be asked to present at the health facility for routine HIV testing. Routine linkage to confirmatory testing and ART initiation will be conducted.
  Arms: Aim 2: Index HIVST

SUMMARY:
This study comprises two trials to evaluate the feasibility and cost-effectiveness of HIV self-testing strategies compared to standard of care among clients in outpatient departments (OPD; Aim 1) and the sexual partners of HIV-positive clients (index testing; Aim 2).

Aim 1 will be a cluster-randomized trial in 15 clusters (high-burden health facilities) in Malawi. We will enroll 6,000 adult OPD clients (15 years or older) to test the feasibility and cost-effectiveness of facility-based HIV self-testing (HIVST) for OPD clients.

Aim 2 will be an individually-randomized trial in 3 high-burden health facilities in Malawi. We will enroll 500 adult HIV-positive clients (15 years or older) to test the feasibility and cost-effectiveness of index HIVST among partners of HIV-positive clients.

DETAILED DESCRIPTION:
The study includes two unblinded trials to evaluate the feasibility and cost-effectiveness of HIVST strategies among adults in Malawi.

Aim 1 will test the feasibility and cost-effectiveness of facility-based HIVST in OPD sites in Malawi. It will be an unblinded cluster-randomized trial and include three arms: 1) standard of care for provider-initiated testing and counseling (PITC); (2) optimized standard of care for PITC; and (3) facility-based HIVST while clients wait for routine OPD services. The standard of care arm will receive no intervention. The optimized standard of care arm will receive training and support for implementing the Malawi guidelines for PITC and morning testing. OPD clients in the facility HIVST arm will receive a HIVST demonstration and distribution, followed by uses of HIVST and private spaces for kit interpretation before receiving routine OPD services. Participants may present their self-test results to their provider, who will refer them for confirmatory HIV testing and routine ART initiation (if positive). That same day, participants from all arms will complete a brief survey upon exiting the clinic. Survey and medical record data will be compared across arms to determine whether facility HIVST is superior in regard to number of individuals tested for HIV, cost-effectiveness, number of HIV-positive individuals identified, and linkage rates for those who identify as HIV-positive.

Aim 2 will test the feasibility and cost-effectiveness of index HIVST for the sexual partners of HIV-positive clients. It will be an unblinded individually-randomized trial and include two arms: 1) standard of care partner referral slips for testing; and 2) HIVST. The standard of care arm will receive no intervention for partner notification and referral. HIV-positive clients in the HIVST arm will receive a HIVST demonstration and distribution, with instructions to give the HIVST kit to their sexual partner. Participants will be given one HIVST for each of their sexual partners who has an unknown HIV status or who tested HIV-negative more than six months prior (up to 3 HIVST kits distributed). Participants (index clients) will be given instructions on how their partner can complete the self-test and how to refer their partner(s) to care if they receive a positive result from the self-test. All participants (standard of care and HIVST arms) will complete a brief survey at the beginning of the intervention and a 4-week follow-up survey to assess primary and secondary outcomes. Medical chart reviews will be conducted for all partners reported to test HIV-positive in order to assess ART initiation rates. Survey and medical record data will be compared across arms to determine whether index HIVST is superior in regard to number of partners tested for HIV, cost-effectiveness, number of HIV-positive individuals identified, and linkage rates for those who identify as HIV-positive.

ELIGIBILITY:
Inclusion Criteria:

* 15 years or older
* Willing and able to provide informed consent
* Being seen for OPD services at the time of the study (Aim 1)
* HIV-positive (Aim 2)
* Have at least one sex partner in the catchment area with an unknown HIV status at the time of study enrollment (Aim 2)

Exclusion Criteria:

* Currently enrolled in the INTERVAL study
* Guardians attending clinics with OPD clients (Aim 1)
* History of intimate partner violence in the past 12 months (Aim 2)
* Fear of intimate partner violence as a consequence of participating in the study (Aim 2)

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6369 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Dovel, PhD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- Partners in Hope, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dovel K, Balakasi K, Phiri K, Shaba F, Offorjebe OA, Gupta SK, Wong V, Lungu E, Nichols BE, Masina T, Worku A, Hoffman R, Nyirenda M. Effect of index HIV self-testing for sexual partners of clients enrolled in antiretroviral therapy (ART) programs in Malawi: A randomized controlled trial. PLoS Med. 2023 Aug 4;20(8):e1004270. doi: 10.1371/journal.pmed.1004270. eCollection 2023 Aug. PMID 37540649
- [Derived] Mphande M, Campbell P, Hoffman RM, Phiri K, Nyirenda M, Gupta SK, Wong V, Dovel K. Barriers and facilitators to facility HIV self-testing in outpatient settings in Malawi: a qualitative study. BMC Public Health. 2021 Dec 2;21(1):2200. doi: 10.1186/s12889-021-12213-6. PMID 34856958
- [Derived] Dovel K, Shaba F, Offorjebe OA, Balakasi K, Nyirenda M, Phiri K, Gupta SK, Wong V, Tseng CH, Nichols BE, Cele R, Lungu E, Masina T, Coates TJ, Hoffman RM. Effect of facility-based HIV self-testing on uptake of testing among outpatients in Malawi: a cluster-randomised trial. Lancet Glob Health. 2020 Feb;8(2):e276-e287. doi: 10.1016/S2214-109X(19)30534-0. PMID 31981557
- [Derived] Dovel K, Shaba F, Nyirenda M, Offorjebe OA, Balakasi K, Phiri K, Nichols B, Tseng CH, Bardon A, Ngona K, Hoffman R. Evaluating the integration of HIV self-testing into low-resource health systems: study protocol for a cluster-randomized control trial from EQUIP Innovations. Trials. 2018 Sep 17;19(1):498. doi: 10.1186/s13063-018-2878-y. PMID 30223874

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited during routine health services at participating facilities. For Aim 1, participants were recruited from September 18, 2017 - February 19, 2018. For Aim 2, participants were recruited from March 21, 2018 - June 13, 2018.
Units Other Than Participants: Facilities
Period: Overall Study
Arm/Group | AIm 1: Standard of Care | Aim 1: Optimized Standard of Care | Aim 1: Facility HIVST | Aim 2: Standard of Care | Aim 2: Index HIVST
Started | 1951; 5 Facilities | 1837; 5 Facilities | 2097; 5 Facilities | 135; 1 Facilities | 349; 2 Facilities
Completed | 1951; 5 Facilities | 1837; 5 Facilities | 2097; 5 Facilities | 107; 1 Facilities | 258; 2 Facilities
Not Completed | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities | 28; 0 Facilities | 91; 0 Facilities
Not completed — Lost to Follow-up | 0 | 0 | 0 | 28 | 91

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIm 1: Standard of Care | Aim 1: Optimized Standard of Care | Aim 1: Facility HIVST | Aim 2: Standard of Care | Aim 2: Index HIVST | Total
Number analyzed (Participants) | 1951 | 1837 | 2097 | 135 | 349 | 6369
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 280 | 223 | 264 | 5 | 6 | 778
  Between 18 and 65 years | 1594 | 1543 | 1800 | 126 | 337 | 5400
  >=65 years | 77 | 71 | 33 | 4 | 6 | 191
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [26 to 35] | 36 [25 to 48] | 35 [28 to 44] | 35 [29 to 45] | 36 [28 to 43] | 35 [27 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1327 | 1002 | 1304 | 105 | 266 | 4004
  Male | 624 | 835 | 793 | 30 | 83 | 2365
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1951 | 1837 | 2097 | 135 | 349 | 6369
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 1951 | 1837 | 2097 | 135 | 349 | 6369
Tested for HIV ≥3months ago [Count of Participants; unit: Participants] | 625 | 508 | 320 | 0 | 0 | 1453

OUTCOME MEASURES:

1. Primary Outcome: Aim 1: Proportion of Adult OPD Clients Tested for HIV
Description: Same day HIV testing among OPD clients, measured by self-reports from OPD clients
Time Frame: 1 day
Population: Descriptive statistics (mean, standard deviation, median, inter-quartile range, and frequency distribution) were generated for the demographic and clinical information to characterize the study population.
Measure: Count of Participants; unit: Participants
Arm/Group | AIm 1: Standard of Care | Aim 1: Optimized Standard of Care | Aim 1: Facility HIVST | Aim 2: Standard of Care | Aim 2: Index HIVST
Number analyzed (Participants) | 1951 | 1837 | 2097 | 0 | 0
Participants | 1951 | 1837 | 2097 |  |

2. Primary Outcome: Aim 2: Proportion of Sexual Partners Tested for HIV
Description: HIV testing among sexual partners of HIV-positive clients within 4-weeks of study enrollment, measured by secondary reports from HIV-positive clients
Time Frame: 4-weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIm 1: Standard of Care | Aim 1: Optimized Standard of Care | Aim 1: Facility HIVST | Aim 2: Standard of Care | Aim 2: Index HIVST
Number analyzed (Participants) | 0 | 0 | 0 | 107 | 258
Participants |  |  |  | 107 | 258

3. Secondary Outcome: Aim 1: HIV-positivity Rate
Description: HIV-positivity rate among OPD clients, measured by self-report
Time Frame: Same 1 day as enrollment (measuring HIV testing before clients leave the OPD clinic that day)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIm 1: Standard of Care | Aim 1: Optimized Standard of Care | Aim 1: Facility HIVST | Aim 2: Standard of Care | Aim 2: Index HIVST
Number analyzed (Participants) | 1951 | 1837 | 2097 | 0 | 0
Participants | 1951 | 1837 | 2097 |  |

4. Secondary Outcome: Aim 1: ART Initiation Among OPD Clients Tested HIV-positive
Description: ART initiation within 3-months after being identified as HIV-positive within the study, measured by medical chart reviews of all Partners in Hope supported health facilities in participating districts
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIm 1: Standard of Care | Aim 1: Optimized Standard of Care | Aim 1: Facility HIVST | Aim 2: Standard of Care | Aim 2: Index HIVST
Number analyzed (Participants) | 1951 | 1837 | 2097 | 0 | 0
Participants | 1951 | 1837 | 2097 |  |

5. Secondary Outcome: Aim 1: Presence of Non-serious Adverse Events
Description: Presence of adverse events due to the HIV testing intervention, including coercion to test, share test results, and unwanted status disclosure, measured by self-report on the day the intervention was delivered.
Time Frame: as enrollment (measuring adverse events that occurred at the OPD clinic that 1 day)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIm 1: Standard of Care | Aim 1: Optimized Standard of Care | Aim 1: Facility HIVST | Aim 2: Standard of Care | Aim 2: Index HIVST
Number analyzed (Participants) | 1951 | 1837 | 2097 | 0 | 0
Participants | 1951 | 1837 | 2097 |  |

6. Secondary Outcome: Aim 1: Cost Per Person Initiated ART
Description: Total cost per arm (including human resources, testing, training, equipment, facility over head, staff, and testing supplies) / total number of individual initiated ART by each arm, respectively. All costs in 2017 US$. Cost calculations do not include cost of ART. Cost data in each study group were derived from a health care perspective using micro-costing methods using the HIV Counselling and Testing costing tool developed by the Health Economics and Epidemiology Research Office in South Africa. All costs are reported in 2017 US$. We use mean cost per ART initiate. Standard deviation is not included due to the nature of calculating a 'production cost'- or the total cost incurred per the respective number of outcomes.
Time Frame: 3 months
Population: Total testing-related costs per person initiated on ART were calculated by study group.
Measure: Mean (Standard Deviation); unit: US dollar
Arm/Group | Aim 1: Standard of Care | Aim 1: Optimized Standard of Care | Aim 1: Facility HIVST
Number analyzed (Participants) | 248 | 261 | 1063
US dollar | 121.02 (NA) — Standard deviation not calculated due to nature of calculating a 'production cost'- or the total cost incurred per the respective number of outcomes | 156.27 (NA) — Standard deviation not calculated due to nature of calculating a 'production cost'- or the total cost incurred per the respective number of outcomes | 279.18 (NA) — Standard deviation not calculated due to nature of calculating a 'production cost'- or the total cost incurred per the respective number of outcomes

7. Secondary Outcome: Aim 2: HIV-positivity Rates Among Sexual Partners Tested for HIV
Description: HIV-positivity rate measured by secondary report by the HIV-positive client
Time Frame: 4-weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIm 1: Standard of Care | Aim 1: Optimized Standard of Care | Aim 1: Facility HIVST | Aim 2: Standard of Care | Aim 2: Index HIVST
Number analyzed (Participants) | 0 | 0 | 0 | 107 | 258
Participants |  |  |  | 107 | 258

8. Secondary Outcome: Aim 2: ART Initiation Among Sexual Partners Tested HIV-positive
Description: as for outcome 4
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIm 1: Standard of Care | Aim 1: Optimized Standard of Care | Aim 1: Facility HIVST | Aim 2: Standard of Care | Aim 2: Index HIVST
Number analyzed (Participants) | 0 | 0 | 0 | 107 | 258
Participants |  |  |  | 107 | 258

9. Secondary Outcome: Aim 2: Presence of Non-serious Adverse Events
Description: Presence of adverse events due to the HIV testing intervention, including coercion to test, share test results, unwanted status disclosure, and interpersonal violence measured by self-report by the HIV-positive client
Time Frame: 4-weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIm 1: Standard of Care | Aim 1: Optimized Standard of Care | Aim 1: Facility HIVST | Aim 2: Standard of Care | Aim 2: Index HIVST
Number analyzed (Participants) | 0 | 0 | 0 | 107 | 258
Participants |  |  |  | 107 | 258

10. Secondary Outcome: Aim 2: Cost Per Person Tested HIV-Positive
Description: Total cost per arm (including human resources, testing, training, equipment, facility over head, staff, and testing supplies) / total number of individual tested HIV-positive by each arm, respectively. All costs in 2017 US$. Cost calculations include all costs associated with HIV testing. Cost data in each study group were derived from a health care perspective using micro-costing methods using the HIV Counselling and Testing costing tool developed by the Health Economics and Epidemiology Research Office in South Africa. All costs are reported in 2017 US$. We use mean cost per HIV-positive individual identified. Standard deviation is not included due to the nature of calculating a 'production cost'- or the total cost incurred per the respective number of outcomes.
Time Frame: 1 month
Population: Arms in Aim 1 not included in this outcome.
Measure: Mean (Standard Deviation); unit: US dollar
Arm/Group | Aim 2: Standard of Care | Aim 2: Index HIVST
Number analyzed (Participants) | 107 | 258
US dollar | 14.9 (NA) — Standard deviation not calculated due to nature of calculating a 'production cost'- or the total cost incurred per the respective number of outcomes | 16.11 (NA) — Standard deviation not calculated due to nature of calculating a 'production cost'- or the total cost incurred per the respective number of outcomes

11. Secondary Outcome: Aim 2: Cost Per Person Initiated ART
Description: as for outcome 6
Time Frame: 3 month
Population: Arms in Aim 1 not included in this outcome
Measure: Mean (Standard Deviation); unit: US dollar
Arm/Group | Aim 2: Standard of Care | Aim 2: Index HIVST
Number analyzed (Participants) | 107 | 258
US dollar | 16.11 (NA) — Standard deviation is not included due to the nature of calculating a 'production cost'- or the total cost | 68.27 (NA) — Standard deviation is not included due to the nature of calculating a 'production cost'- or the total cost

ADVERSE EVENTS:
Time Frame: For Aim 1 (Facility-based HIVST at OPD), adverse events were collected the same day as study enrollment, intervention, and assessment of outcomes. For Aim 2 (Index HIVST), adverse events were collected 4-weeks after study enrollment and delivery of the intervention (HIVST).
Description: For Aim 1, adverse events included (1) coercion to test or share test results; and (2) unwanted status disclosure. Data were collected from follow-up surveys with OPD clients enrolled in the study.
  For Aim 2, adverse events included (1) coercion to test or share test results; (2) unwanted status disclosure; (3) intimate personal violence to the HIV-positive client; and (4) end of the romantic relationship. Data were collected from follow-up surveys with ART clients enrolled in the study.
Arm/Group | AIm 1: Standard of Care | Aim 1: Optimized Standard of Care | Aim 1: Facility HIVST | Aim 2: Standard of Care | Aim 2: Index HIVST
All-Cause Mortality (participants affected / at risk) | 0/1951 | 0/1837 | 0/2097 | 0/107 | 0/258
Serious Adverse Events (participants affected / at risk) | 0/1951 | 0/1837 | 0/2097 | 0/107 | 0/258
Other Adverse Events (participants affected / at risk) | 0/1951 | 0/1837 | 0/2097 | 0/107 | 0/258

LIMITATIONS AND CAVEATS:
Aim 2 data rely on secondary reports from ART clients regarding HIV testing and test results for their sexual partner. Secondary reports may be bias, however, are findings are similar to other HIVST studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT03271307/Prot_SAP_000.pdf